CLINICAL TRIAL: NCT06705738
Title: The Effect of Combination of Mediterranean Diet and Oleocanthal in Patients with Mild Cognitive Impairment
Acronym: MeDi-SUPOL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Greek Alzheimer's Association and Related Disorders (Other); University of Glasgow (Other); World Olive Center for Health (Unknown)
Responsible Party: Principal Investigator, Magda Tsolaki, Emeritus Professor Tsolaki Magdalini, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AUTh
Record Dates: First submitted 2024-11-08; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Mediterranean diet; Western type diet; Olive oil polyphenols; Oleocanthal; Mild cognitive impairment; Alzheimer disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The overall design of the study will be a randomized 4-arm parallel controlled clinical trial, single-blinded for the dietary intervention (MeDi and Western diet) and double-blinded for the intervention (SUPOL and placebo).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study will be single-blinded for the neuropsychological assessment evaluators regarding the dietary intervention and double-blinded for the participants and the neuropsychological assessment evaluators regarding the SUPOL intervention to minimise selection bias.
  The PI and the SUPOL supplier will be blinded to SUPOL administration for the proper conduct of this clinical study. If the PI deems medically necessary to reveal the participant's SUPOL or placebo allocation by breaking the blind, every possible effort must be made to keep participants and evaluators blinded until the end of intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1st group (Experimental): 50 participants will follow the MeDi pattern and will receive SUPOL for 12 months.
  Interventions: Dietary Supplement: SUPOL; Other: Dietary Pattern: MeDi
- 2nd group (Placebo Comparator): 50 participants will follow the MeDi pattern and will receive Placebo capsules for 12 months.
  Interventions: Other: Dietary Pattern: MeDi
- 3rd group (Active Comparator): 50 participants will follow the Western diet pattern and will receive SUPOL for 12 months.
  Interventions: Dietary Supplement: SUPOL
- 4th group (No Intervention): 50 participants will follow the Western diet pattern and will receive Placebo capsules for 12 months.

INTERVENTIONS:
Dietary Supplement: SUPOL — Supplement containing Olive Oil Polyphenol with the main substance being Oleocanthal (SUPOL), 2 capsules twice a day (4 capsules total) for 12 months.
  Arms: 1st group; 3rd group
Other: Dietary Pattern: MeDi — Adherance to Mediterranean dietary pattern to be followed for 12 months.
  Arms: 1st group; 2nd group

SUMMARY:
BACKGROUND: Mild cognitive impairment (MCI) constitutes a form of preclinical dementia and characterizes a cognitive decline that exceeds what is expected for one's age and education status, but at the same time does not fulfill the criteria for dementia. MCI is considered a prodromal stage of Alzheimer's disease (AD) and the progression to this neurodegenerative disease, renders the patients heavily dependent on their relatives and the society, which creates a huge psychological and financial burden, since no effective treatment exists for MCI and AD to this day. Mediterranean diet (MeDi) displays beneficial effects on the cognitive function of both healthy individuals and cognitive impaired patients. High Phenolic Early Harvest Extra Virgin Olive Oil (HP-EH-EVOO) is a natural product that contains high concentrations of the substance Oleocanthal (OLC), while at the same time it has been shown to exert beneficial properties on the cognitive function of cognitive impaired individuals, as well as on the slowing down of the decline of cognitive function.

AIM: The main hypothesis that will be evaluated is whether the combined approach of the MeDi pattern and the concurrent intervention with the administration in a capsule form of the supplement containing olive oil polyphenols with the main substance being Oleocanthal (SUPOL), could constitute a considerable strategy of management of MCI patients.

Study Type: Investigational Study Design, Allocantion: Randomized Intervention Model, Parallel Assignment Masking: Single Blind (Outcome Assessor - Investigator) on Diet, Double Blind (Subject, Outcome Assessor - Investigator) on Supplement, Primary Purpose: Prevention.

DETAILED DESCRIPTION:
OBJECTIVE OF THE TRIAL: To evaluate the efficacy of the combined approach of the MeDi pattern and the concurrent SUPOL compared to the Western diet pattern in combination with placebo on the change in cognition and function in subjects with MCI.

STUDY DESIGN: The design will be a randomized parallel controlled clinical trial, single-blinded for the dietary pattern and double-blinded for the intervention.

PARTICIPANTS: They will be divided into 4 groups of 50 (n=200): 1st group following MeDi and receiving SUPOL, 2nd group following MeDi and receiving Placebo, 3rd group following Western type diet (Western diet) and receiving SUPOL and 4th group following Western diet and receiving Placebo.

DURATION: The duration of the combined intervention will be 12 months and the neuropsychological and laboratory evaluation of the participants will take place at baseline and upon the completion of the 1-year combined intervention. A follow-up assessment visit will be perfomed after 6 monts. The total study duration will be 18 months.

LOCATION: The study will be conducted in Thessaloniki and will recruit patients having diagnosed with MCI from the outpatient clinic 1st Neurological Clinic of the General University Hospital "AHEPA" (AHEPA) and the Greek Association of Alzheimer's Disease and Related Disorders (Alzheimer Hellas).

SCREENING - RANDOMIZATION - BASELINE (Visit 1): Patient eligibility will be determined during Visit 1. A protocol eligibility form will be completed for each patient and reviewed by the Principal Investigator (PI) approval prior to participation in the study. If eligibility is reached, baseline assessments, as well as randomization for group allocation will take place.

ELIGIBILITY:
Inclusion criteria:

Participants are eligible to be included in this study only if all the following criteria apply:

* Men or women,
* 60 to 85 years of age inclusive, at the time of signing the informed consent form (ICF).
* Mini-Mental State Examination (MMSE) score of 26-28 at Screening (Visit 1).
* Montreal Cognitive Assessment (MoCA) score of 20-26 at Visit 1.
* MRI scan evaluation at Visit 1.
* CSF biomarkers evaluation at Visit 1.
* Adequate knowledge and understanding of the Greek language, as well as adequate literacy, vision and hearing for neuropsychological testing in the opinion of the Principal Investigator (PI) at the time of screening.
* They are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical conditions

* Significant neurological diseases that affect the central nervous system other than MCI, that may affect cognition ability to complete the study, including but not limited to, other dementias, serious infection of the brain, Parkinson's disease (PD), Multiple sclerosis (MS), multiple concussions, epilepsy or recurrent seizures.
* Ongoing serious or unstable illnesses, including cardiovascular, hepatic, renal, gastroenterological, respiratory, endocrinologic, psychiatric, immunologic, hema-tologic diseases and other conditions that, in the PI's opinion, could interfere with the analyses in this study or has a life expectancy of less than 24 months.
* History of cancer within the last 5 years, with exception of non-metastatic basal and/or squamous cell carcinoma of the skin, in situ cervical cancer, nonprogressive prostate cancer, other cancers with low risk of recurrence or spread.
* Participants with any current primary psychiatric diagnosis, if in the judgement of the PI for the psychiatric disorder or symptom is likely to confound interpretation of the combined approach effect, affect cognitive assessment or affect the partici-pant's ability to complete the study. Participants with history of schizophrenia or other chronic psychosis are excluded.
* In the judgement of the PI, participants are actively suicidal and therefore deemed to be at significant risk of suicide.
* History of alcohol or drug abuse disorder (except tobacco use disorder) within 2 years before Visit 1.
* History of clinically significant multiple or severe drug allergies, significant atopy or severe post-treatment hypersensitivity reactions (including but not limited to erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis and/or exfoliative dermatitis).
* Patient has undergone surgical operation of the gastrointestinal tract (GI tract) that led to removal of a functional part of the GI tract, length shortage of the GI tract and change of the GI tract morphology.

Imaging, Vital Signs, Laboratory Tests and Physical Examinations

* Any clinically important abnormality at Visit 1, as determined by the PI, in physical or neurological examination, vital signs or clinical laboratory test results, that could be detrimental to the participant, could compromise the study or show evidence of other etiologies for MCI.
* MRI which shows evidence of significant abnormality that would suggest another potential etiology for MCI or a clinically significant finding that may impact the participant's ability to safely participate in the study.
* Have any contraindications for MRI, including claustrophobia or the presence of contraindicated metal (ferromagnetic) implants/cardiac pacemaker.
* Poor venous access.
* Evidence of a relevant neurological disorder other than MCI at Visit 1, including but not limited to PD, Lewy body disease, frontotemporal dementia of any type, Huntington's disease, amyotrophic lateral sclerosis, MS, systemic lupus erythematosus, progressive supranuclear palsy, neurosyphilis, HIV, learning disability, intellectual disability, hypoxic cerebral damage, or significant head trauma with loss of consciousness that led to persistent cognitive deficits.
* Evidence of a clinically relevant or unstable psychiatric disorder, based on Diag-nostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria, including schizophrenia or other psychotic disorder, or bipolar disorder. A subject with a history of major depression who has not had an episode in the last 24 months before the day of screening and is considered in remission or in the case that depression is controlled with treatment can be included in the trial per inves-tigator's judgement.
* Imminent risk of self-harm, based on clinical interview and responses on the Columbia Suicide Severity Rating Scale (C-SSRS) or of harm to self or others in the opinion of the PI.

Prior or Concomitant Therapy

* Known allergies to EVOO, OLC, Oleacein (OLE), Oleuropein Aglycon (OLA), Ligstroside Aglycon (LIG), Tyrosol (TYR), Hydroxytyrosol (HT) or any other components of the formulation.
* Contraindications in following a MeDi or Western diet pattern and are not willing to adhere to the abovementioned nutritional lifestyles.
* Consumption of high-dose nutritional supplements.
* Long-term antibiotic therapy.
* Regular consumption of probiotics.
* Regular intake of enriched commercial probiotic foods.

Prior or Concurrent Clinical Study Experience

* Currently enrolled in any other interventional clinical trial involving an investigational medicinal product (IMP) or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Participated, within the last 30 days in a clinical trial involving an IMP. If the precious IMP is scientifically or medically incompatible with this study and has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed prior to Visit 1 (participation in observational studies may be permitted upon review or the observational study protocol and approved by the PI).
* Previously completed or withdrawn from this study or received SUPOL in any prior investigational study. (This exclusion criterion does not apply to participants who are allowed to rescreen before randomization in this study).

Other exclusions

* Investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Currently OMPHAX SA (OMPHAX) employees or employees of third-party organizations (TPOs) involved in study which requires exclusion of their employees or have relatives or partners who are OMPHAX employees or are employees of TPOs involved in a study which requires exclusion of their employees.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
ADAS-Cog - Measurement to Assess the Severity of Cognitive Impairment | Baseline (Day 1) to 12 months
  Alzheimer's Disease Assessment Scale - Cognitive Subscale - 13 (ADAS-Cog-13) neuropsychological assessment scale scores ranges from 0 to 85, with greater scores showing a more significant cognitive impairment
MMSE - Measurement to Assess and Evaluate Cogntive Function | Baseline (Day 1) to 12 months
  Mini-Mental State Examination (MMSE) score ranges range from 0 to 30 and individuals will lower MMSE scores show greater cognitive impairment

SECONDARY OUTCOMES:
MoCA - Measurement to Assess Cognitive Abilities | Baseline (Day 1) to 12 months
  Montreal Cognitive Assessment (MoCA) total score ranges from 0 to 30 and lower scores indicating greater impairment
ADCS-ADL-MCI - Measurement to Assess and Evaluate the Performance in Different Activities of Daily Living | Baseline (Day 1) to 12 months
  Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale for Mild Cognitive Impairment (ADCS-ADL-MCI) MCI scale score ranges from 0 to 53, with poorer scores representing a more significant cognitive impairment
CDR-SB - Measurement to Assess the Severity of the Disease and the Progression of the Disease | Baseline (Day 1) to 12 months
  Clinical Dementia Rating Sum of Boxes (CDR-SB) total score ranges from 0 to 18, with greater scores corresponding to more significant impairment
CDR - Measurement of Time to Progression to Dementia | Baseline (Day 1) to 12 months
  Clinical Dementia Rating (CDR) global score ranges from 0 to 3, with the higher score corrisponding to severe dementia and the time to progression to dementia will be measured in weeks (unit)
GDS - Measurement to Identify Depression in the Elderly | Baseline (Day 1) to 12 months
  Geriatric Depression Scale (GDS) total score ranges from 0 to 30, with the classification of severity to be: (a) normal 0-9, (b) mild depression 10-19 and (c) severe depression 20-30
C-SSRS - Measurement to Determine the Potential Risk for Suicide | Baseline (Day 1) to 12 months
  Columbia - Suicide Severity Rating Scale (C-SSRS) score ranges from 2 to 25, with the higher number indicating more intense suicidal ideation
TEAEs - Measurment of Number of Treatment Emergent Adverse Events | Baseline (Day 1) to 12 months
  Number of treatment emergent adverse events (TEAEs) are measured in number of events from baseline
Measurement of Change in the Vital Signs | Baseline (Day 1) to 12 months
  Number of participants with change from baseline in blood pressure (measured in mmHg) will be assessed
Measurement of Change in the Vital Signs | Baseline (Day 1) to 12 months
  Number of participants with change in pulse rate (heart beats per minute) will be assessed
Measurement of Change in Physical Examination | Baseline (Day 1) to 12 months
  Number of participants with change from baseline in physical examination will be evaluated
Measurement of Change in Neurological Examination | Baseline (Day 1) to 12 months
  Number of participants with change from baseline on neurological examination will be evaluated
Measurment of Change in Clinical Laboratory Tests | Baseline (Day 1) to 12 months
  Number of participants with change from baseline in biochemical test will be evaluated
Measurement of Change in Clinical Laboratory Tests | Baseline (Day 1) to 12 months
  Number of participants with change from baseline in haematological test wiil be evaluated

OTHER OUTCOMES:
Measurment of Change in Plasma Aβ1-42 | Baseline (Day 1) to 12 months
  Change in mean values of beta-amyloid 1-42 protein (Aβ1-42) plasma concentration
Measurment of Change in Plasma Aβ1-40 | Baseline (Day 1) to 12 months
  Change in mean values of beta-amyloid 1-40 protein (Aβ1-40) plasma concentration
Measurement of Change in the Aβ1-42/Aβ1-40 Plasma Ratio | Baseline (Day 1) to 12 months
  Change in the Amyloid-β1-42/Amyloid-β1-40 (Aβ1-42/Aβ1-40) ration in plasma levels
Measurment of Change in Plasma pTau-181 | Baseline (Day 1) to 12 months
  Change in mean values of phosphorylated Tau-181 protein (pTau-181) plasma concentration
Measurment of Change in Plasma pTau-217 | Baseline (Day 1) to 12 months
  Change in mean values of phosphorylated Tau-217 protein (pTau-217) plasma concentration
Measurment of Change in Plasma GFAP | Baseline (Day 1) to 12 months
  Change in mean values of Glial Fibrillary Acidic Protein (GFAP) plasma concentration
Measurement of Change in Plasma IL-1β | Baseline (Day 1) to 12 months
  Change in mean value of Inteleukin-1β (IL-1β) plasma levels
Measurement of Change in Plasma IL-6 | Baseline (Day 1) to 12 months
  Change in mean value of Inteleukin-6 (IL-6) plasma levels
Measurement of Change in Plasma CRP | Baseline (Day 1) to 12 months
  Change in mean value of C-Reactive Protein (CRP) plasma levels
Measurement of Change in Gut Microbiota Composition | Baseline (Day 1) to 12 months
  Change in gut microbiome alpha-diversity (α-diversity) and beta-diversity (β-diversity)
Measurment of Change in Gut Microbiome Metabolites | Baseline (Day 1) to 12 months
  Change in the gut microbiome short chain fatty acids (SCFAs) and medium chain fatty acids (MCFAs) concentration

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - "AHEPA" General University Hospital of Thessaloniki, Thessaloniki, Thessaloniki
  - Greek Association of Alzheimer's Disease and Related Disorders, Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: No
No plans to share data with other researchers